CLINICAL TRIAL: NCT01281657
Title: A Long Term, Multicenter, Non-interventional, Observational Study Monitoring Long-term Safety and Effectiveness of Fingolimod 0.5 mg in Patients With Multiple Sclerosis Who Have Participated in the Fingolimod Clinical Development Program
Brief Title: Long Term Study of Fingolimod in MS Patients From the FTY Clinical Program
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CFTY720D2399E1
Record Dates: First submitted 2011-01-19; First posted 2011-01-24 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Sclerosis
Keywords: Fingolimod; FTY720; Relapsing forms of multiple sclerosis; Multiple sclerosis; MS; Safety; Efficacy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prescribed fingolimod 0.5 mg/day
  Interventions: Drug: fingolimod

INTERVENTIONS:
Drug: fingolimod

SUMMARY:
The purpose of this observational study is to collect long-term data on safety and effectiveness of fingolimod, particularly including clinical disease and patient outcome related parameters such as relapse and disability, in patients who have participated in prior trials within the fingolimod clinical development program. Furthermore, this study explores the incidence of selected safety related outcomes of fingolimod treatment during follow-up visits within the context of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed fingolimod as part of their routine medical care
* Patients who have participated in a prior fingolimod clinical trials

Exclusion Criteria:

* Restrictions regarding the use of fingolimod while pregnant or nursing in accordance with the local prescribing label
* Any patient who has prematurely discontinued from the previous fingolimod trial

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing forms of MS who have participated in previous fingolimod trials and now taking commercially available fingolimod as part of routine medical care
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Long-term safety data in patients with relapsing forms of multiple sclerosis who have participated in clinical trials with fingolimod and who are now taking prescribed fingolimod under the conditions of routine medical practice | Throughout the entirety of the study up to a maximum of 8 years

SECONDARY OUTCOMES:
Long-term effectiveness data, particularly including clinical disease and patient outcome related parameters such as relapse and disability | Throughout the entirety of the study up to a maximum of 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- United States (42):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - The Research & Education Inst. of Alta Bates Summit Med. Grp, Berkeley, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - University of California San Francisco, San Francisco, California
  - Yale Multiple Sclerosis Center, New Haven, Connecticut
  - Georgetown University/Lombardi Cancer Center, Washington D.C., District of Columbia
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - University of Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - AMO Corporation, Tallahassee, Florida
  - MS Center of Vero Beach, Vero Beach, Florida
  - South Suburban Neurology, Flossmoor, Illinois
  - Neurologic Associates, LTD, Palos Heights, Illinois
  - Mercy Ruan Neurology Clinic Res Ct., Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mid America Neuroscience Institute, Lenexa, Kansas
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins MS Center, Baltimore, Maryland
  - Caritas St. Elizabeth's Hospital, Boston, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Spectrum Health Medical Group, Neurology, Grand Rapids, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - The MS Center for Innovation in Care, St Louis, Missouri
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Island Neurological Associates, Plainview, New York
  - SUNY - Stony Brook University, Stony Brook, New York
  - University of Toledo Health Science Campus, Toledo, Ohio
  - MS Center of Oklahoma, Oklahoma City, Oklahoma
  - Neurological Associates of Tulsa, Inc, Tulsa, Oklahoma
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jerfferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Medical School, Houston, Texas
  - Integra Clinical Research, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - Dean Foundation, Madison, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (14):
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Nepean, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan